CLINICAL TRIAL: NCT07380230
Title: Efficacy and Safety of Qibei Jiedu Formula Versus Placebo in Preventing and Managing Acute Radiation Dermatitis in Breast Cancer Patients: A Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Qibei Jiedu Formula for Preventing and Managing Acute Radiation Dermatitis in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LI FENG (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, LI FENG, Director and Chief Physician, Department of Traditional Chinese Medicine, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 25/468-5594
Record Dates: First submitted 2026-01-19; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Radiation Dermatitis; Traditional Chinese Medicine (TCM); Breast Cancer
Keywords: Acute radiation dermatitis; Integrated Traditional Chinese and Western Medicine; Breast Cancer; Traditional Chinese Medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Standard Basic Treatment:
  All patients will receive guideline-based hypofractionated radiotherapy (40-50 Gy/15 fractions) and routine skin care (e.g., hydrogel dressings or creams) determined by the treating physician. The specific products and usage must be documented in the CRF and maintained as stable as possible after enrollment.
  Add-on Intervention:
  Patients will be randomly assigned to receive either Qibei Jiedu Formula or its simulator (5% of the original formula dosage), taken from the first day of radiotherapy. One decocted dose (divided into two 100-mL bags) is taken twice daily for 21 days (synchronized with radiotherapy).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Standard basic treatment + Qibei Jiedu Formula
  Interventions: Drug: Standard Basic Treatment Combined with Qibei Jiedu Formula
- Control Group (Experimental): Standard basic treatment + Qibei Jiedu Formula simulator (containing 5% of the original formula dosage)
  Interventions: Drug: Standard Basic Treatment Combined with Qibei Jiedu Formula simulator

INTERVENTIONS:
Drug: Standard Basic Treatment Combined with Qibei Jiedu Formula — Participants will commence administration of either the Qibei Jiedu Formula on the first day of radiotherapy. The daily regimen consists of one decocted dose, divided into two sealed bags (specification: 100 mL per bag). One bag is to be taken orally twice daily (morning and evening) for a continuous period of 3 weeks (21 days, synchronized with the radiotherapy course).
  Arms: Treatment Group
Drug: Standard Basic Treatment Combined with Qibei Jiedu Formula simulator — Participants will begin taking either the simulator (containing 5% of the original formula dosage) on the first day of radiotherapy. The daily dose consists of one formula unit, decocted and divided into two bags of medicinal liquid (specification: 100 mL per bag). Participants are to take one bag per dose, twice daily (morning and evening), for a continuous period of 3 weeks (21 days, synchronized with the radiotherapy course).
  Arms: Control Group

SUMMARY:
1. To evaluate the preventive and therapeutic effects of Qibei Jiedu Formula on acute radiation dermatitis in breast cancer patients, including the incidence of grade 2 or higher radiation dermatitis, wound healing time, and symptom relief.
2. To observe the safety profile of Qibei Jiedu Formula.
3. To investigate the potential role of Qibei Jiedu Formula in improving patients' quality of life.
4. To explore the potential mechanism of action of Qibei Jiedu Formula in preventing and treating acute radiation dermatitis in breast cancer patients through exploratory indicators such as inflammatory cytokines and skin microbiota.
5. This study is a small-scale exploratory clinical trial. It aims to collect preliminary efficacy and safety data from 60 participants to assess the "add-on effect" of Qibei Jiedu Formula on top of "standard basic care". The results are intended for estimating effect sizes and generating hypotheses to inform future large-scale studies, not for drawing definitive conclusions.

DETAILED DESCRIPTION:
Acute Radiation Dermatitis (ARD) following breast cancer radiotherapy has an incidence rate as high as 95%, with grade 3 or higher dermatitis leading to unplanned radiotherapy interruption in 15-20% of patients. This not only compromises treatment efficacy but also significantly impairs patients' quality of life. Current conventional Western medical management primarily relies on corticosteroids and moisturizers, yet faces limitations in efficacy and notable side effects. Developed based on the Fuzheng Quyu Jiedu (Strengthening Vital Qi, Removing Stasis, and Detoxifying) theory, the Qibei Jiedu Formula has shown promising anti-inflammatory, antipruritic, and wound-healing effects in preliminary clinical observations.

Led by Professor Feng Li's team from the Cancer Hospital of the Chinese Academy of Medical Sciences, this project adopts a multicenter, randomized, double-blind, placebo-controlled clinical trial design. It plans to enroll 60 breast cancer patients scheduled for radiotherapy to systematically evaluate the clinical efficacy and safety of Qibei Jiedu Formula in preventing and treating ARD. The study aims to provide high-level evidence-based medical data for the integrated Chinese and Western medicine prevention and management of ARD. Furthermore, it seeks to establish a safer and more effective treatment regimen, thereby reducing unplanned radiotherapy interruptions and improving oncologic outcomes. The findings are expected to offer an evidence-based rationale for the TCM-based prevention and treatment of radiation dermatitis, provide a new option for clinical practice, and contribute positively to enhancing the quality of life of cancer patients, holding significant social value.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed unilateral stage I-III non-inflammatory breast cancer, having undergone breast-conserving surgery or modified radical mastectomy, and having received or planned to receive standard adjuvant therapy according to current clinical guidelines.
* Scheduled to receive postoperative adjuvant radiotherapy using a hypofractionated regimen (40-50 Gy/15 fractions) as recommended by the NCCN Breast Cancer Guidelines and the CSCO Breast Cancer Diagnosis and Treatment Guidelines (2024 Edition).
* Meeting the TCM diagnostic criteria for the syndrome of Qi-Yin Deficiency with Blood Stasis and Toxin Accumulation.
* Karnofsky Performance Status (KPS) score ≥70.
* Age ≥18 years, female.
* Voluntarily participating in the study and providing written informed consent.

Exclusion Criteria:

* Presence of grade 4 radiation dermatitis requiring urgent intervention at enrollment or during the study.
* Prior radiotherapy to the breast or chest within the past 3 months.
* Any skin condition that may interfere with the assessment of radiation dermatitis, such as active infection, atopic dermatitis, psoriasis, vitiligo, active collagen vascular disease (e.g., scleroderma, lupus erythematosus), or other known autoimmune disorders significantly altering skin appearance or physiological response.
* Pre-existing grade ≥2 hepatic/renal dysfunction or hematological toxicity (according to CTCAE v5.0 criteria) before treatment.
* Concurrent participation in other clinical trials or concurrent use of other Chinese herbal preparations.
* Unstable mental status or inability to cooperate with the study procedures.
* Pregnant or lactating patients.
* Known allergy to any component of the herbal formula used in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥2 Acute Radiation Dermatitis | During treatment (Day 7, Day 14, Day 17, Day 21) and 1 month after treatment (Day 49)
  The proportion of participants who develop Grade 2 or higher acute radiation dermatitis during radiotherapy and within 1 month after completion of radiotherapy, as assessed and confirmed by investigators according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Time to Onset of Grade 2 Acute Radiation Dermatitis | During treatment (Day 7, Day 14, Day 17, Day 21) and 1 month after treatment (Day 49)
  Time from the start of radiotherapy to the first occurrence of Grade 2 acute radiation dermatitis, as confirmed by investigators according to CTCAE v5.0.
Time to Wound Healing of Radiation Dermatitis | During treatment (Day 7, Day 14, Day 17, Day 21) and 1 month after treatment (Day 49)
  Time from the first documented occurrence of Grade 2 or 3 acute radiation dermatitis to recovery to less than Grade 2 (Grade 0 or 1), as assessed according to CTCAE v5.0 and the Guidelines for Clinical Research of New Chinese Medicines.
Severity of Radiation Dermatitis Symptoms Assessed by RISRAS | During treatment (Day 7, Day 14, Day 17, Day 21) and 1 month after treatment (Day 49)
  Severity of radiation-induced skin reactions assessed using the Radiation-Induced Skin Reaction Assessment Scale (RISRAS).
  RISRAS is a composite scale consisting of:a patient-reported symptom score (pain, itching, burning, and impact on daily activities), and a clinician-rated skin reaction score.
  Scale Range and Interpretation： Total score range: 0 to 36 Higher scores indicate more severe radiation-induced skin reactions
Quality of Life Assessed by EORTC QLQ-BR23 | Baseline, during treatment (Day 14 and Day 21), and 1 month after treatment (Day 49)
  Quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer Module (EORTC QLQ-BR23).
  Scale Range and Interpretation Scores are linearly transformed to a scale of 0 to 100 Higher scores indicate better quality of life or higher symptom burden, depending on the specific subscale, according to the EORTC scoring manual
Quality of Life Assessed by Dermatology Life Quality Index (DLQI) | Baseline, during treatment (Day 14 and Day 21), and 1 month after treatment (Day 49)
  Dermatology-related quality of life assessed using the Dermatology Life Quality Index (DLQI).
  Scale Range and Interpretation Total score range: 0 to 30 Higher scores indicate greater impairment of dermatology-related quality of life
Traditional Chinese Medicine (TCM) Syndrome Score | Baseline, during treatment (Day 14 and Day 21), and 1 month after treatment (Day 49)
  Severity of Traditional Chinese Medicine (TCM) syndrome assessed using a composite TCM syndrome score scale developed according to the Guidelines for Clinical Research of New Chinese Medicines (2002 edition), the Guidelines for Diagnosis and Treatment of Malignant Tumors in Traditional Chinese Medicine, and External Treatment of Traditional Chinese Medicine.
  The scale evaluates TCM-related symptoms including fatigue, chest tightness and shortness of breath, heat sensations in the palms and soles, dry mouth and throat, localized pain, skin changes, fever with sweating, irritability and insomnia, lip and nail color changes, subcutaneous ecchymosis, dark urine, and constipation.
  Treatment efficacy is evaluated based on changes in the total TCM syndrome score from baseline at different assessment time points.
  Scale Range and Interpretation Total score range: 0 to 54 Higher scores indicate more severe TCM syndrome symptoms
Skin Colorimetric Changes Assessed by Skin Reflectance Spectrophotometry (SRS) | During treatment (Day 7, Day 14, Day 17, Day 21) and 1 month after treatment (Day 49)
  Skin color changes of radiation dermatitis assessed using skin reflectance spectrophotometry with a validated colorimeter. Measurements are performed on the irradiated breast skin, with three readings averaged per site. Skin color is quantified using the CIE L*a*b* color space, and changes from baseline (ΔL*, Δa*, Δb*) are analyzed. Lower ΔL* values indicate increased pigmentation, and higher Δa* values indicate increased erythema severity. Δb* is analyzed as a secondary parameter. Measurements of the contralateral breast are performed at baseline and at the end of radiotherapy to control for systemic skin color changes.

OTHER OUTCOMES:
Blood Inflammatory Levels | At baseline and at the end of treatment (Day 21).
  A 5-mL sample of venous blood was collected from the median cubital vein of each patient, stored in a serum separator tube, and analyzed for inflammatory marker levels using enzyme-linked immunosorbent assay (ELISA).
Skin Microbiota Analysis | At baseline and at the end of treatment (Day 21).
  Samples were collected by swabbing a 5 cm × 5 cm area along the central axis of the radiation field and its border, using non-irradiated skin 2 cm outside the field edge as a control. A sterile cotton swab was used to swab the target area, which was divided into four rectangular sub-areas from top to bottom. The swab tip was kept in firm contact with the skin and moved back and forth at least five times in each sub-area. After swabbing each sub-area, the swab was rotated 90° before proceeding to the next to ensure maximal microbial collection over the entire swab head. After collection, the swab was immediately placed in preservation solution. Skin microbiota analysis was performed using 16S rRNA gene sequencing.
Lymphocyte Subset Analysis | At baseline and at the end of treatment (Day 21).
  A 5-mL venous blood sample was collected from the median cubital vein of each patient, stored in an EDTA-anticoagulated tube, and analyzed for peripheral blood lymphocyte subset distribution by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmeel LC, Koch D, Schmeel FC, Bucheler B, Leitzen C, Mahlmann B, Kunze D, Heimann M, Bruser D, Abramian AV, Schoroth F, Mudder T, Rohner F, Garbe S, Baumert BG, Schild HH, Wilhelm-Buchstab TM. Hydrofilm Polyurethane Films Reduce Radiation Dermatitis Severity in Hypofractionated Whole-Breast Irradiation: An Objective, Intra-Patient Randomized Dual-Center Assessment. Polymers (Basel). 2019 Dec 16;11(12):2112. doi: 10.3390/polym11122112. PMID 31888185
- [Background] Bohner AMC, Koch D, Schmeel FC, Rohner F, Schoroth F, Sarria GR, Abramian AV, Baumert BG, Giordano FA, Schmeel LC. Objective Evaluation of Risk Factors for Radiation Dermatitis in Whole-Breast Irradiation Using the Spectrophotometric L*a*b Color-Space. Cancers (Basel). 2020 Aug 28;12(9):2444. doi: 10.3390/cancers12092444. PMID 32872216
- [Background] Dejonckheere CS, Layer JP, Sarria GR, Wiegreffe S, Glasmacher AR, Nour Y, Scafa D, Mudder T, Anzbock T, Giordano FA, Stope MB, Schmeel LC, Gkika E. Non-invasive physical plasma for preventing radiation dermatitis in breast cancer: study protocol for a phase 3 randomised double-blind placebo-controlled trial (NIPP-RD III). Trials. 2025 Mar 19;26(1):97. doi: 10.1186/s13063-025-08806-w. PMID 40108640
- [Background] Tang Y, Zhou Y, Li HJ. Advances in mesenchymal stem cell exosomes: a review. Stem Cell Res Ther. 2021 Jan 19;12(1):71. doi: 10.1186/s13287-021-02138-7. PMID 33468232
- [Background] Wickenheisser VA, Zywot EM, Rabjohns EM, Lee HH, Lawrence DS, Tarrant TK. Laser Light Therapy in Inflammatory, Musculoskeletal, and Autoimmune Disease. Curr Allergy Asthma Rep. 2019 Jul 2;19(8):37. doi: 10.1007/s11882-019-0869-z. PMID 31267251
- [Background] Hong JP, Lee SW, Song SY, Ahn SD, Shin SS, Choi EK, Kim JH. Recombinant human epidermal growth factor treatment of radiation-induced severe oral mucositis in patients with head and neck malignancies. Eur J Cancer Care (Engl). 2009 Nov;18(6):636-41. doi: 10.1111/j.1365-2354.2008.00971.x. Epub 2009 Apr 23. PMID 19456848
- [Background] Liu C, Wei J, Wang X, Zhao Q, Lv J, Tan Z, Xin Y, Jiang X. Radiation-induced skin reactions: oxidative damage mechanism and antioxidant protection. Front Cell Dev Biol. 2024 Oct 9;12:1480571. doi: 10.3389/fcell.2024.1480571. eCollection 2024. PMID 39450273
- [Background] Rube CE, Freyter BM, Tewary G, Roemer K, Hecht M, Rube C. Radiation Dermatitis: Radiation-Induced Effects on the Structural and Immunological Barrier Function of the Epidermis. Int J Mol Sci. 2024 Mar 15;25(6):3320. doi: 10.3390/ijms25063320. PMID 38542294
- [Background] Xie Y, Wang Q, Hu T, Chen R, Wang J, Chang H, Cheng J. Risk Factors Related to Acute Radiation Dermatitis in Breast Cancer Patients After Radiotherapy: A Systematic Review and Meta-Analysis. Front Oncol. 2021 Nov 29;11:738851. doi: 10.3389/fonc.2021.738851. eCollection 2021. PMID 34912704
- [Background] Han B, Zheng R, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2022. J Natl Cancer Cent. 2024 Feb 2;4(1):47-53. doi: 10.1016/j.jncc.2024.01.006. eCollection 2024 Mar. PMID 39036382
- [Background] Giaquinto AN, Sung H, Miller KD, Kramer JL, Newman LA, Minihan A, Jemal A, Siegel RL. Breast Cancer Statistics, 2022. CA Cancer J Clin. 2022 Nov;72(6):524-541. doi: 10.3322/caac.21754. Epub 2022 Oct 3. PMID 36190501

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT07380230/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT07380230/ICF_001.pdf